CLINICAL TRIAL: NCT00094120
Title: Safety and Efficacy of MSI-1256F (Squalamine Lactate) in Combination With Verteporfin in Patients With "Wet" Age-Related Macular Degeneration (AMD)
Brief Title: MSI-1256F (Squalamine Lactate) in Combination With Verteporfin in Patients With "Wet" Age-Related Macular Degeneration (AMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Genaera Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSI-1256F-208
Record Dates: First submitted 2004-10-11; First posted 2004-10-14 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2007-11

CONDITIONS: Macular Degeneration
Keywords: Age-Related Macular Degeneration - Wet Type
MeSH Terms: conditions — Macular Degeneration | interventions — squalamine lactate

INTERVENTIONS:
Drug: MSI-1256F (Squalamine Lactate)

SUMMARY:
Age-Related Macular Degeneration (AMD) is a degenerative disease of the retina that causes a progressive loss of central vision. AMD is the leading cause of legal blindness among adults age 50 or older in the Western world. AMD presents in two different types - "dry" and the more severe "wet" form. Wet AMD is caused by the growth of abnormal blood vessels in the macula.

Squalamine lactate is an investigational drug that may prevent the growth of these abnormal blood vessels. This study will test the safety and efficacy of Squalamine when administered with verteporfin therapy in patients with "wet" AMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of "wet" age-related macular degeneration

Exclusion Criteria:

* Prior treatment for "wet" age-related macular degeneration

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Genaera Corporation, Plymouth Meeting, Pennsylvania, United States